CLINICAL TRIAL: NCT07260266
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Postoperative Opioid Consumption in Patients Undergoing Major Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Clinical Professor, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-LP-778
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous vagus nerve stimulation(taVNS) (Active Comparator): Patients received taVNS treatment immediately upon entering the AICU, with sessions occurring every 2 hours. A specialized taVNS stimulator device was used, and the left ear was cleaned with an alcohol swab or wet tissue before inserting an earplug with electrode contacts into the left ear, ensuring a snug fit. A second earplug was inserted into the right ear. The stimulation parameters were set as follows: continuous wave, frequency 20 Hz, pulse width 200 μs. Each treatment session lasted for 30 minutes.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation
- Sham-stimulation (Placebo Comparator): The treatment protocol was identical to that of the taVNS group. Electrodes were placed on the left auricle. After the device was activated, it either did not deliver any current or only emitted a brief sub-threshold current to simulate the sensation of device activation, without producing continuous neural stimulation.
  Interventions: Device: Sham Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — Patients received taVNS treatment immediately upon entering the AICU, with sessions occurring every 2 hours. A specialized taVNS stimulator device was used, and the left auricle was cleaned with an alcohol swab or wet tissue before inserting an earplug with electrode contacts into the left ear, ensuring a snug fit. A second earplug was inserted into the right ear. The stimulation parameters were set as follows: continuous wave, frequency of 20 Hz, and pulse width of 200 μs. Each treatment session lasted for 30 minutes.
  Arms: transcutaneous vagus nerve stimulation(taVNS)
Device: Sham Transcutaneous auricular vagus nerve stimulation — The treatment protocol was identical to that of the taVNS group. Electrodes were placed on the left auricle. After the device was turned on, it either did not output any current or only delivered a brief sub-threshold current to simulate the sensation of the device being activated, without producing continuous neural stimulation.
  Arms: Sham-stimulation

SUMMARY:
This study aims to design a prospective, double-blind, randomized controlled trial to compare the effects of transcutaneous auricular vagus nerve stimulation (taVNS) on postoperative visceral pain in patients undergoing major abdominal surgery. Participants will be randomly assigned to receive either taVNS or sham stimulation. The total consumption of opioids and other analgesics within 24 hours post-surgery in the AICU will be recorded, along with follow-up assessments of pain scores and quality of recovery scores (Qor-15) at 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years, regardless of gender
* ASA physical status classification I-III
* Scheduled for elective major abdominal surgery under general anesthesia, with postoperative admission to the AICU for monitoring
* Anticipated duration of stay in the AICU is approximately 24 hours

Exclusion Criteria:

* History of vagus nerve-related diseases (such as vasovagal syncope);
* Severe arrhythmias or implanted electronic devices such as pacemakers;
* Skin lesions, infections, or deformities at the site of external ear stimulation;
* Long-term preoperative use of opioid medications or sedatives;
* Allergy to study-related medications;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Total consumption of opioids | within 24 hours postoperatively.
  Total consumption of opioids (morphine equivalent) within 24 hours postoperatively.

SECONDARY OUTCOMES:
sleep quality score | Postoperative first-night
  Postoperative first-night sleep quality score (Richards-Campbell Sleep Questionnaire, RCSQ); the score ranges from 0 to 150, with higher scores indicating better sleep quality.
Quality of Recovery Score | 24 Hours Post-Operatively
  Quality of Recovery Score (QoR-15) at 24 Hours Post-Operatively;The score ranges from 0 to 150 points, with higher scores indicating better postoperative recovery quality.
Adverse events associated with taVNS | 24 Hours Postoperatively
  Adverse events associated with taVNS (local skin irritation, dizziness, tinnitus, etc.);
The incidence of opioid-related complications | within 24 hours post-surgery
  The incidence of opioid-related complications (such as respiratory depression, nausea and vomiting, and intestinal paralysis) within 24 hours post-surgery.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol